CLINICAL TRIAL: NCT04542343
Title: Multilevel, Multidisciplinary, Faith-Based Participatory Interventions to Reduce COVID-19 Related-Risks Among Underserved African Americans
Brief Title: COVID-19 Risk Reduction Among African American Parishioners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: COVID19Church; 5U54MD007598-15 (NIH)
Record Dates: First submitted 2020-09-03; First posted 2020-09-09 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections | interventions — Health Resources

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Risk Reduction of COVID-19 Among African American Parishioners (Experimental): This arm will implement "one group pretest-posttest" design to improve COVID associated health outcomes of AA older parishioners in collaboration with trained young church-based health educators.
  Interventions: Behavioral: Change in knowledge, motivation, skills, resources

INTERVENTIONS:
Behavioral: Change in knowledge, motivation, skills, resources — Provide/enhance knowledge, modify attitudes, motivate and provide skills and resources to reduce COVID-19 related risk and challenges.

SUMMARY:
African American adults, specifically those managing chronic disease and social isolation, are one of the most vulnerable groups susceptible to COVID-19. This intervention involves a multi-disciplinary and culturally sensitive approach to address two major COVID-19 related challenges in this population. First, this program collaborates with predominantly African American churches to implement Federal and State guidelines aimed at preventing outbreaks of COVID-19 at faith-based gatherings. Second, this program trains church-based health advisors to help African American older parishioners manage their chronic health conditions and reduce psychological distress during the pandemic.

DETAILED DESCRIPTION:
To jointly implement and evaluate a telehealth-based, multidisciplinary, culturally-sensitive intervention with 265 AA older parishioners: (i) To mitigate the negative impact of COVID-19 on the management of chronic health conditions, and (ii) to reduce healthcare avoidance behaviors and psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* African American older adults aged 55 years with a chronic medical condition or 65years and older
* Have at least one risk factor for COVID-19

Exclusion Criteria:

* Resident of care facility
* Cognitive deficit (identified by short version of mini-mental instrument)
* Does not self-identify as African American and/or Black
* Under the age of 55years
* Unable to speak and/or read English

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Bazargan, PhD, Principal Investigator — Charles R. Drew University of Medicine & Science
Locations (1):
- Charles R. Drew University of Medicine & Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Aim 1: Faith-based Leadership: This arm involves a series of workshops aimed at enhancing faith-based leaders' understanding and communication skills regarding COVID-19 prevention and health safety measures. The training focuses on enabling leaders to effectively disseminate critical COVID-19 information within their communities.
- Aim 2: COVID-19 Health Ambassadors: This group is part of a community outreach program where selected individuals from partnered faith-based organizations are trained to act as health ambassadors. The intervention includes comprehensive training on COVID-19 health practices, with an emphasis on support for chronic disease management, medication adherence, psychosocial support and, compliance with personal and public safety measures.
- Aim 3: Older African American Adults: This intervention is designed specifically for older African American adults, focusing on enhancing their ability to manage chronic conditions and navigate health-related challenges during the COVID-19 pandemic. The program includes educational workshops, personalized health management plans, and community support systems to assist older parishioners in maintaining their health and safety led by trained health ambassadors. Key aspects of the intervention include training on how to safely visit healthcare providers, manage medication refills, and understand the importance of preventative measures against COVID-19.
Period: Overall Study
Arm/Group | Aim 1: Faith-based Leadership | Aim 2: COVID-19 Health Ambassadors | Aim 3: Older African American Adults
Started | 17 | 46 | 152
Completed | 10 | 19 | 110
Not Completed | 7 | 27 | 42

BASELINE CHARACTERISTICS:
Population: AIM1: Faith-based Leadership The arm consists of recruited faith-based leaders who play a pivotal role in community guidance and influence.
  Aim 2: COVID-19 Health Ambassadors Participants were recruited from various faith-based organizations showing interest in health advocacy.
  AIM 3: Older African American Adults The participants in this group are older adultswho are particularly vulnerable to COVID-19 and often face multiple challenges in managing chronic health conditions.
Groups:
- Aim 1: Faith-based Leadership: This arm targets faith-based leaders and involves a series of workshops aimed at enhancing their understanding and communication skills regarding COVID-19 prevention and health safety measures. The training focuses on enabling leaders to effectively disseminate critical COVID-19 information within their communities.
- Aim 2: COVID-19 Health Ambassadors: This group is part of the project's community outreach where selected individuals are trained to act as lay health advisors (health ambassadors). The intervention includes comprehensive training on COVID-19 health practices, with an emphasis on chronic disease management.
- Aim 3: Older African American Adults: This intervention is tailored specifically for older adults within the church community, focusing on enhancing their ability to manage chronic conditions and navigate health-related challenges during the COVID-19 pandemic. The program includes educational workshops and personalized health management plans facilitated and supported by trained health ambassadors. These ambassadors directly assist older parishioners in understanding and applying preventive measures against COVID-19, safely managing medication refills, and ensuring safe visits to healthcare providers.
- Total: Total of all reporting groups
Arm/Group | Aim 1: Faith-based Leadership | Aim 2: COVID-19 Health Ambassadors | Aim 3: Older African American Adults | Total
Number analyzed (Participants) | 10 | 19 | 110 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 10 | 29 | 43
  >=65 years | 6 | 9 | 81 | 96
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 15 | 77 | 94
  Male | 8 | 4 | 33 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 19 | 110 | 139
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Ability to Implement COVID-19 Health Guidelines Among African American Churches in South Los Angeles 3 Months After Workshop
Description: This measure evaluates the readiness of African American church leaders in South Los Angeles to reopen their churches according to Federal and State COVID-19 guidelines. It specifically assesses their confidence and ability to implement safety protocols learned during the workshops, using the "Church Reopening Preparedness" construct of the Church Leaders' Pandemic Outreach & Preparedness Scale (CLOPS) [Cronbach's alpha of 0.97]. This construct measures effectiveness on a Likert scale from 1 (strongly disagree) to 5 (strongly agree), reflecting how well leaders apply these protocols to ensure a safe worship environment. Higher Scores indicate effective readiness to implement safety measures. Lower Scores suggest areas where further training or planning is needed. Positive numbers indicate increases in preparedness to reopen faith-based organizations.
Time Frame: 3 months. The assessments were conducted immediately before the workshop (baseline) and repeated three months after to measure changes in preparedness.
Measure: Mean (95% Confidence Interval); unit: score on a scale of 1-5
Arm/Group | Aim 1: Faith-based Leadership
Number analyzed (Participants) | 10
score on a scale of 1-5 | 3.00000 [2.24600 to 3.75400]
Statistical Analysis 1: Comparison: Aim 1: Faith-based Leadership; Test type: Other; p < 0.01, t-test, 2 sided; Mean Difference (Net) = 3.00000, 95% CI 2-sided [2.24600 to 3.75400]

2. Primary Outcome: Mean Change in COVID-19 Knowledge Among Faith-based Leaders After Educational Workshop
Description: Church Leaders' Pandemic Outreach & Preparedness Scale (CLOPS) is designed to assess the effectiveness of COVID-19 workshops in changing the preparedness of church leaders to reopen churches and to deepen their knowledge about COVID-19 (Cronbach's alpha of 0.97) . Positive mean differences indicate increases in preparedness to reopen these faith-based organizations. The general COVID-19 knowledge enhancement construct measures the increase in participants' understanding of COVID-19, including its transmission and preventive measures on a Likert scale from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate an enhanced knowledge of COVID-19 (better outcome). Lower scores suggest gaps in workshop content or participant comprehension (worse outcome).
Time Frame: 3 days from the start of the workshops (baseline) to completion of workshop training sessions.
Population: Church leaders who participated in the pre and post-assessment of the COVID-19 training workshops on adoption of COVID-19 public health guidelines
Measure: Mean (95% Confidence Interval); unit: score on a scale of 1-5
Groups:
- Aim 1: Faith-Based Leadership: Evaluation of the educational effectiveness of the COVID-19 training workshops for faith-based leaders on adoption of guidelines
Arm/Group | Aim 1: Faith-Based Leadership
Number analyzed (Participants) | 10
score on a scale of 1-5 | -3.30000 [-4.256785 to -2.343215]
Statistical Analysis 1: Comparison: Aim 1: Faith-Based Leadership; Test type: Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -3.30000, 95% CI 2-sided [-4.256785 to -2.343215]

3. Primary Outcome: Number of Faith-based COVID-19 Health Ambassadors Who Attended at Least 2 Out of the 3-Day Training Workshops
Description: The outcome measure was primarily determined by the count of health ambassadors' attendance in a minimum of two out of three training sessions (each session held daily). These 3-day sessions encompassed interactive discussions and informal knowledge assessments designed to ensure comprehension and retention of critical COVID-19 information. The informal assessments were diverse, including group discussions where participants articulated preventive measures against COVID-19, role-playing to exemplify how they would convey complex health information to various community demographics, particularly older adults with underlying health conditions, and impromptu Q&A segments aimed at evaluating participants' understanding of essential topics and rectifying any misconceptions immediately.
Time Frame: 3 days from the start of the workshops (baseline) to completion of workshop training sessions.
Population: Number of participants who attended at least two out of the three day training workshops.
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 2: COVID-19 Health Ambassadors
Number analyzed (Participants) | 19
Participants | 19

4. Primary Outcome: Mean Change in Preparedness for COVID-19 Testing, Vaccination, and Health Promotion by Health Ambassadors After Training Workshop
Description: This outcome measure assesses the effectiveness of COVID-19 workshops in changing ambassadors' preparedness across five key constructs, as defined in CLOPS, including discussing infection risks, changing attitudes towards testing, boosting motivation for vaccination, convincing vaccine-hesitant individuals, and supporting older parishioners in managing chronic conditions amid the pandemic. Each construct is evaluated using a Likert scale from 1 to 5, where higher scores reflect a high level of readiness and effectiveness in demonstrating strong persuasive abilities, communication skills, and a capacity to support healthcare needs. Conversely, lower scores pinpoint areas requiring enhanced training, additional resources, or improved strategies. The total score is the sum of all sub-scale scores and ranges from 5 to 25. A negative mean difference between combined construct scores indicates an increase in the post-workshop scores compared to the pre-workshop scores.
Time Frame: 3 days from the start of the workshops (baseline) to completion of workshop training sessions.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aim 2: COVID-19 Health Ambassadors
Number analyzed (Participants) | 19
score on a scale | -16.4 [-19.96 to -12.64]

5. Primary Outcome: Total Number of Older Adult Parishioners Who Filled/Refilled at Least One of Their Prescription(s) After 6 Months Intervention With Support From a Health Ambassador
Description: This measure assesses the total number of participants who successfully filled/refilled at least one medication at the end of the intervention. Older adult participants, with the help of health ambassadors, self-reported whenever they picked up a medication fill/refill from their pharmacy. Only participants with outstanding prescriptions were required to report. By this, the outcome seeks to evaluate the effectiveness of the intervention in enhancing medication management among older adults, particularly in navigating health-related challenges during the COVID-19 pandemic.
Time Frame: 6 months. The end of the intervention was marked by 6 months after the first scheduled meeting (baseline) between the health ambassador and older adult parishioners.
Population: Total number of participants who filled/refilled at least one of their prescription(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 3: Older African American Adults
Number analyzed (Participants) | 110
Participants | 80

6. Primary Outcome: Total Number of Older Adult Parishioners Who Received at Least One COVID-19 Vaccine After 6 Months Intervention With Support From a Health Ambassador
Description: Assessing the number of participants who had received at least one additional COVID-19 vaccine by the end of the intervention period with the aid of a health ambassador
Time Frame: 6 months. The end of the intervention was marked by 6 months after the first scheduled meeting (baseline) between the health ambassador and church members.
Measure: Count of Participants; unit: Participants
Arm/Group | Aim 3: Older African American Adults
Number analyzed (Participants) | 110
Participants | 107

7. Primary Outcome: Mean Change in Healthcare Utilization Among Older Adult Parishioners After 6 Months Intervention With Support From a Health Ambassador
Description: This measure examines the delay in healthcare utilization among study participants with an emphasis on understanding the effects of interventions aimed at reducing barriers to accessing primary care, specialty services, dental care, and medication fills. To quantify these delays, a scale called the Healthcare Utilization Delay Scale was created, incorporating four distinct constructs: delay in getting prescriptions filled or refilled, visiting primary care providers, receiving dental care, and visiting specialty services. Scores on the scale are from 0 (no delay in any service) to 4 (delay in all measured services). Higher scores indicate more delays in healthcare utilization, representing a worse outcome, whereas lower scores suggest fewer delays, indicating better access to healthcare services. A negative mean difference indicates reduction in healthcare utilization delay among parishioners (calculated as post- minus pre-intervention scores).
Time Frame: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aim 3: Older African American Adults
Number analyzed (Participants) | 110
score on a scale | -0.21818 [-0.36828 to -0.06809]
Statistical Analysis 1: Comparison: Aim 3: Older African American Adults; Test type: Other; p < 0.01, t-test, 2 sided; Mean Difference (Net) = -0.21818, 95% CI 2-sided [-0.36828 to -0.06809]

8. Primary Outcome: Mean Change in COVID-19 Knowledge Among Parishioners After 6 Months Intervention With Support From a Health Ambassador
Description: This outcome measure assesses the effectiveness of an intervention by health ambassadors designed to increase COVID-19 knowledge among older adult parishioners using a newly developed 19-item scale - COVID-19 Knowledge Scale (Cronbach alpha = 0.87).Each item on the scale assesses participants' understanding of key aspects of COVID-19, such as transmission methods, symptoms, prevention strategies, and treatment options, with responses recorded as binary (1 = correct or 0 = incorrect). The total knowledge score for each participant is derived by averaging the scores across all items, with potential scores ranging from 0 to 1 (actual average scores ranged from 0.10 to 1.0). Higher average scores on this scale indicate a better understanding of COVID-19, and improvements are reflected by a positive mean difference in scores before and after the intervention (calculated as post- minus pre-intervention scores).
Time Frame: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aim 3: Older African American Adults
Number analyzed (Participants) | 110
score on a scale | 0.05623 [0.00459 to 0.10788]
Statistical Analysis 1: Comparison: Aim 3: Older African American Adults; Test type: Other; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 0.05623, 95% CI 2-sided [0.00459 to 0.10788], Standard Error of Mean 0.026

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Aim 1: Faith-based Leadership | Aim 2: COVID-19 Health Ambassadors | Aim 3: Older African American Adults
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/46 | 0/152
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/46 | 0/152
Other Adverse Events (participants affected / at risk) | 0/17 | 0/46 | 0/152

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT04542343/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT04542343/ICF_001.pdf